CLINICAL TRIAL: NCT05857371
Title: Safety and Potential Effect of Innovative Treatment by Adjuvant Injection of Stromal Vascular Fraction From Autologous Adipose Tissue of URethral Stenosis With Endoscopic Urethrotomy: Randomized Controlled Trial
Brief Title: Safety and Potential Effect of Innovative Treatment by Adjuvant Injection of Stromal Vascular Fraction From Autologous Adipose Tissue of URethral Stenosis With Endoscopic Urethrotomy
Acronym: SURF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCAPHM18_0020_1; 2022-002175-11 (EudraCT Number)
Record Dates: First submitted 2023-02-03; First posted 2023-05-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Urethral Stenosis
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): The surgeon trained to lipoaspiration procedure will perform lipoaspiration for the ADSVF cryopreservation under local anesthesia with sedation.
  The patients of the control group benefices to urethrotomy (standard care) under general anesthesia. The surgical surgical technique necessitates performing three incisions with a cold endoscopic knife in the stenosis to obtain enlargement of urethral lumen on the length of the fibrosis at 3, 9 and 12 o' clock.
  For patients randomised in the control group, lippoaspiration will be performed for cryopreservation of the autologous ADSVF and potential second administration of ADSVF in case of UrS recurrency. UrS recurrence or primary failure is defined as a recurrence without a period of post procedure improvement). Recurrence incoming before 21 months post experimental treatment will be treated according to the study in order to have a minimum follow-up of 3 months.
  Interventions: Procedure: lipoaspiration; Procedure: urethrotomy
- Experimental group (Experimental): The surgeon trained to lipoaspiration procedure will perform lipoaspiration for the ADSVF cryopreservation under local anesthesia with sedation.
  The patients of the control group benefices to urethrotomy (standard care) under general anesthesia. The surgical surgical technique necessitates performing three incisions with a cold endoscopic knife in the stenosis to obtain enlargement of urethral lumen on the length of the fibrosis at 3, 9 and 12 o' clock.
  For theses patients -randomised in the experimental group - the experimental cell drug will be customised-made to each patient's lesion and included a dose between 16 and 56 million* viable nucleated cells (VNCs) of fresh or thawed autologous Adipose-derived -Stromal Vascular Fraction, resuspended in saline (0, 9%) - 5% human serum albumin (50 mg/mL) final packaged in 2 to 7 syringes of 1 mL at a concentration of 8 million CNV / mL, individually closed with a tamper-proof Luer Lock cap and labelled to ensure double-blindness.
  Interventions: Procedure: lipoaspiration; Procedure: urethrotomy; Drug: autologous ADSVF administration

INTERVENTIONS:
Procedure: lipoaspiration — The surgeon will perform lipoaspiration under local anesthesia for the ADSVF production.
Procedure: urethrotomy — The urologist will perform an endoscopic urethrotomy (standard care).
Drug: autologous ADSVF administration — ADSVF will be administrated in fibrotic lesion during urethrotomy by the urologist.
  Arms: Experimental group

SUMMARY:
SURF is a randomised controlled, parallel group, single blind phase II study designed to assess the safety and potential efficacy of an innovative therapeutic strategy for urethral stenosis based on adjuvant injection of autologous Adipose-Derived Stromal Vascular Fraction of Adipose Tissue (ADSVF) during endoscopic urethrotomy (standard care).

DETAILED DESCRIPTION:
Urethral stenosis (UrS) is a narrowing of the urethra's caliber. UrS results of ischemic fibrosis of the corpus spongiosum (spongiofibrosis). Fibrosis-induced retraction reduces the size of the urethral lumen. Spongiofibrosis may be due to infections, inflammation, trauma but remains mostly idiopathic.Endo-urethral treatment exposes to a high rate of recurrence (up to 60% depending on the site, length and etiology). The reconstruction treatment is more effective but more complex (use of oral mucosal flap or other substitution tissue, less mastered by the surgical community and more morbid.

The (ADSVF) is an easily accessible source of autologous mesenchymal stem cells. Obtention from lipoaspirates is safe, simple and standardized. Different animal models have demonstrated the pro-healing and anti-fibrotic properties of autologous ADSVF in the urethra corpus cavernous during erectile dysfunction, perineal fistulas during Crohn's disease and systemic sclerosis.

The main objective of this study is to assess the safety and tolerability of ADSVF, as add-on treatment to endoscopic urethrotomy for recurrent bulbar urethral stenosis during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male, aged from 18 to 85 years
* Bulbar urethral stenosis ≤ 3 cm.
* At least one urethral dilatation or urethrotomy for the bulbar stenosis in the past 24 months before diagnosis of stenosis
* Ability to avoid corticoids or immunosuppressive drugs one month after treatment. For any patients with either corticoid or immunosuppressive treatment the physician in charge of this treatment will be contacted and asked to give a written approval for one month cessation of the therapy
* Good general health status according to clinical history and a physical examination
* BMI > 18 to insure adequate access to abdominal or other subcutaneous adipose tissue for adipose tissue harvesting

Exclusion Criteria:

* Urethral stenosis of other location than bulbar
* Urethral stenosis length > 3 cm
* Urethral stenosis on reconstructed penis (transgender, post amputation)
* Prior perineal or pelvic radiotherapy
* Concurrent urinary tract infection without treatment
* Concurrent perineal infection
* Penile cancer < 5 years
* Current or recent history of abnormal, severe, progressive, uncontrolled infectious, hepatic, haematological, gastrointestinal (except CD), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease
* Congenital or acquired immunodeficiencies
* Contraindication to the anaesthetic or surgical procedure
* Corticoids or immunosuppressive drugs > 3 months
* Any active viral infection among the following: HIV, HTLV I and II, VHB, VHC and syphillis
* Administrative restricted rights
* Presence of signs of obstructive voiding symptoms not directly attributable to the stricture at the discretion of the physician
* Diagnosis of untreated and unresolved BPH benign prostatic hyperplasia or BNC bladder neck contracture
* Diagnosis of carcinoma of the urethra, bladder or prostate within the last two (2) years

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identtity
Enrollment: 20 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Baseline intensity and duration of urethral pain | 1 day
  A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain D7 | 7 days
  measured 7 days after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M1 | 1 month
  measured 1 month after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M3 | 3 months
  measured 3 months after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M6 | 24 months
  measured 6 months after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M9 | 9 months
  measured 9 months after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M18 | 18 months
  measured 18 months after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Intensity and duration of urethral pain M24 | 24 months
  measured 24 months after therapeutic administration. A degree of pain can be expected at the tissue sampling site. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institute.
Incidence of urinary infection | 24 months
  measured at baseline (day of inclusion). This adverse event will be collected during clinical examination from blood sample analysis.
Incidence of urniary infection M1 | 1 month
  measured 1 month after therapeutic administration. This adverse event will be collected during clinical examination from blood sample analysis.
Number of patient with urethral bleeding | 1 day
  measured at baseline (day of inclusion). This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding D7 | 7 days
  measured 7 days after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M1 | 1 month
  measured 1 month after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M3 | 3 months
  measured 3 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M6 | 6 months
  measured 6 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M9 | 9 months
  measured 9 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M18 | 18 months
  measured 18 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Number of patient with urethral bleeding M24 | 24 months
  measured 24 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institut.
Presence of urethral perforation with fistula or perineal soft tissue infection D7 | 7 days
  measured 7 days after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institut.
Presence of urethral perforation with fistula or perineal soft tissue infection M1 | 1 month
  measured 1 month after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Presence of urethral perforation with fistula or perineal soft tissue infection M3 | 3 months
  measured 3 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Presence of urethral perforation with fistula or perineal soft tissue infection M6 | 6 months
  measured 6 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Presence of urethral perforation with fistula or perineal soft tissue infection M9 | 9 months
  measured 9 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator. The events intensity will be graded according to the version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE) classification (grade 1 to 5 toxicity) of National Cancer Institut.
Presence of urethral perforation with fistula or perineal soft tissue infection M18 | 18 months
  measured 18 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.
Presence of urethral perforation with fistula or perineal soft tissue infection M24 | 24 months
  measured 24 months after therapeutic administration. This adverse event will be collected during clinical examination from the investigator questioning the patient; or from the patient's unsolicited reporting, as encouraged to do towards the investigator.

SECONDARY OUTCOMES:
USP score | 24 months
  Change from baseline Urinary Symptom Profile (USP) scores at 1, 3, 6, 9, 18 and 24 months. USP scores include 3 different scales :
  * low stream score. Minimum score = 0 ; Maximum score (worse outcome) = 9
  * overactivity score. Minimum score = 0 ; Maximum score (worse outcome) = 21
  * stress incontinence. Minimum score = 0 ; Maximum score (worse outcome) = 9
International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms Module (ICIQ-MLUTS) | 24 months
  Change from baseline ICIQ-MLUTS at 1, 3, 6, 9, 18 and 24 months. Minimum score = 0 ; Maximum score (worse outcome) = 21
Uroflowmetry | 24 months
  Uroflowmetry is a noninvasive test of the voiding phase. It consists in a device which assess urine flow (Q max normal >12ml/s, shape of the curve) and the urinated volume. To be interpreted Uroflowmetry needs to be coupled with a post micturition residual volume mesasure via an automated bladder sonography device. Urinated volume + residual volume known as bladder pre-charge and needs to be higher than 150ml to make the uroflowmetry nterpretable and meaningful.
  Urinary change from baseline will be measured at 1, 3, 6, 9, 18 and 24 months.
Baseline imaging assessment of spongiofibrosis volume with Fat Sat sequences | 24 months
  A magnetic-resonance imaging (MRI) will be performed locally at Screening (baseline), to assess the volume of spongiofibrosis using Sagittal view in T1 Fat Sat after Gadolinium injection.
imaging assessment of spongiofibrosis volume with Fat Sat sequences M1 | 24 months
  A magnetic-resonance imaging (MRI) will be performed locally at M1 to assess the volume of spongiofibrosis using Sagittal view in T1 Fat Sat after Gadolinium injection.
imaging assessment of spongiofibrosis volume with Fat Sat sequences M9 | 24 months
  A magnetic-resonance imaging (MRI) will be performed locally at M9 to assess the volume of spongiofibrosis using Sagittal view in T1 Fat Sat after Gadolinium injection.
Recurrence rate | 24 months
  Recurrence of urethral stenosis (defined as a recurrence without a period of post procedure improvement) will be analyzed at 1, 3, 6,9 18, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIX CREMIEUX, Study Director — ASSISITANCE PUBLIQUE HOPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France